CLINICAL TRIAL: NCT07016282
Title: Simulated and Synthetic Health Data: Improving Clinical Research on Rare Diseases. A Real-World Data Simulation of Autosomal Dominant Polycystic Kidney Disease (ADPKD) Trials. A Retrospective, Observational Study
Acronym: SAILING-ADPKD
Status: Active, not recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: SAILING-ADPKD
Record Dates: First submitted 2025-05-27; First posted 2025-06-11 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: rare diseases; RCTs; Monte Carlo simulation; generative AI; ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Rare Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Real-world data form ADPKD patients: Real-world data from ADPKD-related electronic health records (EHR) stored at the Istituto di Ricerche Farmacologiche Mario Negri IRCCS, primarily based on the ALADIN (NCT00309283) and ALADIN 2 (NCT01377246) studies
- Simulated data: Data based on RWD from the ADPKD patients and derived from predefined statistical models (e.g., normal distribution for continuous variables, binomial distribution for categorical variables).
- Synthetic data: Data generated from the RWD of the ADPKD patients using generative large languages models (LLMs)

SUMMARY:
This is a no-profit, retrospective observational study involving real-world data (RWD), retrieved from ADPKD-related electronic health records stored at Mario Negri Institute IRCCS. RWD will be used to generate simulated and synthetic datasets, using AI tools. RWD and generated data (GD) will be used to conduct three virtual RCTs, which main outcome is change in Total Kidney Volume (TKV). Statistical tests will be performed to assess quality and privacy preservation of GD compared with RWD. GD will be also evaluated in exploratory sample size estimations.

DETAILED DESCRIPTION:
Randomized clinical trials (RCTs) can be regarded as the least biased source of information to address intervention questions. One of the most common problems encountered in clinical trials focused on rare diseases is the difficulty in finding patients and therefore in building trials on sufficiently large population, in order to have more robust data and less methodological distortions. Several stratagems are already in use to deal with these problems, including extended trial duration, repeated outcome measures, patients genetic profiles, surrogate endpoint, multicenter studies. Another approach is to consider other trial designs in addition to parallel-arms design, such as crossover trial, n-of-1 trials, and adaptive trials.

Simulated and synthetic health data can represent new valid approaches to increase the representativeness of the patients, especially in rare diseases field, while reducing costs and time constraints, but also facing the limitations imposed by national and international regulations concerning privacy and data management. Simulation studies are defined as computer experiments that involve creating data by pseudo-random sampling from known probability distributions, based on Monte Carlo method. A promising approach now under development includes synthetic data, defined as artificially generated data with the aim of reproducing the statistical properties of an original dataset, through generative large languages models (LLMs).

Thus, while simulated data rely on known distributions that must be specified in advance, synthetic data are generated by LLMs that learn these distributions from training data, without the need for predefined distributions, offering a significant advantage in flexibility and applicability.

This study aims to find the most suitable tool for generating simulated and synthetic data in rare diseases field, and to compare the fidelity, quality, and privacy preservation of these datasets, derived from real-world ADPKD clinical trial data. Furthermore, a virtual clinical trial will be conducted using these three datasets to assess their validity in replicating real trial outcomes.

Finally, retrieved and generated data will be used to assess new sample size estimations for future clinical trial performed at the Clinical Research Center for Rare Disease "Aldo e Cele Daccò", Istituto di Ricerche Farmacologiche Mario Negri IRCCS, Ranica (BG), Italy.

By using generative AI models, such as Generative Adversarial Networks (GANs), this study aims to overcome challenges related to data poverty and trial design. The results could provide valuable insights into whether synthetic data can be a useful tool for improving clinical trials in rare diseases, making them more efficient and cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) men and women with ADPKD according to Ravine criteria25
* Estimated glomerular filtration rate (eGFR) between 15 and 40 mL/min/1.73 m2 (CKD stage: G3b-G4) or higher (CKD stage: G1-G3a), as calculated by the Modification of Diet in Renal Disease study four variables equation

Exclusion Criteria:

* confounding factors that could affect renal function loss independent of kidney growth and treatment allocation (i.e., diabetes mellitus, urinary protein excretion rate >3 g/24 h)
* Abnormal urinalysis suggestive of concomitant, clinically significant glomerular disease, and urinary tract lithiasis or infection
* Patients with major systemic disease
* Patients unable to provide informed consent
* Pregnant, lactating, or potentially childbearing women without adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from ADPKD patients collected in the form of electronic health records (EHR) stored at the Istituto di Ricerche Farmacologiche Mario Negri IRCCS, primarily based on two completed studies performed at the Mario Negri Institue i.e., the ALADIN Study (NCT00309283) and the ALADIN 2 Study (NCT01377246), which enrolled ADPKD-patients treated either with Octreotide-LAR or placebo.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Changes in total kidney volume (TKV) | At baseline, and immediately after data generation procedure.
  Changes in TKV in mL.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, M.D., Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (2):
- Clinical Research Centre for Rare Diseases Aldo e Cele Daccò, Ranica, BG, Italy
- Department of Global Public Health (GPH), Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bolignano D, Pisano A. Good-quality research in rare diseases: trials and tribulations. Pediatr Nephrol. 2016 Nov;31(11):2017-23. doi: 10.1007/s00467-016-3323-7. Epub 2016 Jan 27. PMID 26817476
- [Background] Halpern SD, Karlawish JH, Berlin JA. The continuing unethical conduct of underpowered clinical trials. JAMA. 2002 Jul 17;288(3):358-62. doi: 10.1001/jama.288.3.358. PMID 12117401
- [Background] Lilford RJ, Thornton JG, Braunholtz D. Clinical trials and rare diseases: a way out of a conundrum. BMJ. 1995 Dec 16;311(7020):1621-5. doi: 10.1136/bmj.311.7020.1621. PMID 8555809
- [Background] Gagne JJ, Thompson L, O'Keefe K, Kesselheim AS. Innovative research methods for studying treatments for rare diseases: methodological review. BMJ. 2014 Nov 24;349:g6802. doi: 10.1136/bmj.g6802. PMID 25422272
- [Background] Shurin S, Krischer J, Groft SC. Clinical trials In BMT: ensuring that rare diseases and rarer therapies are well done. Biol Blood Marrow Transplant. 2012 Jan;18(1 Suppl):S8-11. doi: 10.1016/j.bbmt.2011.10.030. No abstract available. PMID 22226117
- [Background] van der Lee JH, Wesseling J, Tanck MW, Offringa M. Efficient ways exist to obtain the optimal sample size in clinical trials in rare diseases. J Clin Epidemiol. 2008 Apr;61(4):324-30. doi: 10.1016/j.jclinepi.2007.07.008. Epub 2008 Feb 21. PMID 18313556
- [Background] Stone EM. Challenges in genetic testing for clinical trials of inherited and orphan retinal diseases. Retina. 2005 Dec;25(8 Suppl):S72-S73. doi: 10.1097/00006982-200512001-00034. No abstract available. PMID 16374347
- [Background] Buckley BM. Clinical trials of orphan medicines. Lancet. 2008 Jun 14;371(9629):2051-5. doi: 10.1016/S0140-6736(08)60876-4. No abstract available. PMID 18555919
- [Background] Kinder B, McCormack FX. Clinical trials for rare lung diseases: lessons from lymphangioleiomyomatosis. Lymphat Res Biol. 2010 Mar;8(1):71-9. doi: 10.1089/lrb.2009.0027. PMID 20235889
- [Background] Lagakos SW. Clinical trials and rare diseases. N Engl J Med. 2003 Jun 12;348(24):2455-6. doi: 10.1056/NEJMe030024. No abstract available. PMID 12802033
- [Background] Berlin JA. N-of-1 clinical trials should be incorporated into clinical practice. J Clin Epidemiol. 2010 Dec;63(12):1283-4. doi: 10.1016/j.jclinepi.2010.05.006. Epub 2010 Aug 30. PMID 20800449
- [Background] Cerqueira FP, Jesus AMC, Cotrim MD. Adaptive Design: A Review of the Technical, Statistical, and Regulatory Aspects of Implementation in a Clinical Trial. Ther Innov Regul Sci. 2020 Jan;54(1):246-258. doi: 10.1007/s43441-019-00052-y. Epub 2020 Jan 6. PMID 32008232
- [Background] Yoon J, Drumright LN, van der Schaar M. Anonymization Through Data Synthesis Using Generative Adversarial Networks (ADS-GAN). IEEE J Biomed Health Inform. 2020 Aug;24(8):2378-2388. doi: 10.1109/JBHI.2020.2980262. Epub 2020 Mar 12. PMID 32167919
- [Background] Morris TP, White IR, Crowther MJ. Using simulation studies to evaluate statistical methods. Stat Med. 2019 May 20;38(11):2074-2102. doi: 10.1002/sim.8086. Epub 2019 Jan 16. PMID 30652356
- [Background] METROPOLIS N, ULAM S. The Monte Carlo method. J Am Stat Assoc. 1949 Sep;44(247):335-41. doi: 10.1080/01621459.1949.10483310. No abstract available. PMID 18139350
- [Background] Chen RJ, Lu MY, Chen TY, Williamson DFK, Mahmood F. Synthetic data in machine learning for medicine and healthcare. Nat Biomed Eng. 2021 Jun;5(6):493-497. doi: 10.1038/s41551-021-00751-8. PMID 34131324
- [Background] Caroli A, Perico N, Perna A, Antiga L, Brambilla P, Pisani A, Visciano B, Imbriaco M, Messa P, Cerutti R, Dugo M, Cancian L, Buongiorno E, De Pascalis A, Gaspari F, Carrara F, Rubis N, Prandini S, Remuzzi A, Remuzzi G, Ruggenenti P; ALADIN study group. Effect of longacting somatostatin analogue on kidney and cyst growth in autosomal dominant polycystic kidney disease (ALADIN): a randomised, placebo-controlled, multicentre trial. Lancet. 2013 Nov 2;382(9903):1485-95. doi: 10.1016/S0140-6736(13)61407-5. Epub 2013 Aug 21. PMID 23972263
- [Background] Perico N, Ruggenenti P, Perna A, Caroli A, Trillini M, Sironi S, Pisani A, Riccio E, Imbriaco M, Dugo M, Morana G, Granata A, Figuera M, Gaspari F, Carrara F, Rubis N, Villa A, Gamba S, Prandini S, Cortinovis M, Remuzzi A, Remuzzi G; ALADIN 2 Study Group. Octreotide-LAR in later-stage autosomal dominant polycystic kidney disease (ALADIN 2): A randomized, double-blind, placebo-controlled, multicenter trial. PLoS Med. 2019 Apr 5;16(4):e1002777. doi: 10.1371/journal.pmed.1002777. eCollection 2019 Apr. PMID 30951521
- [Background] Cornec-Le Gall E, Alam A, Perrone RD. Autosomal dominant polycystic kidney disease. Lancet. 2019 Mar 2;393(10174):919-935. doi: 10.1016/S0140-6736(18)32782-X. Epub 2019 Feb 25. PMID 30819518
- [Background] Chebib FT, Perrone RD, Chapman AB, Dahl NK, Harris PC, Mrug M, Mustafa RA, Rastogi A, Watnick T, Yu ASL, Torres VE. A Practical Guide for Treatment of Rapidly Progressive ADPKD with Tolvaptan. J Am Soc Nephrol. 2018 Oct;29(10):2458-2470. doi: 10.1681/ASN.2018060590. Epub 2018 Sep 18. PMID 30228150
- [Background] Ravine D, Gibson RN, Walker RG, Sheffield LJ, Kincaid-Smith P, Danks DM. Evaluation of ultrasonographic diagnostic criteria for autosomal dominant polycystic kidney disease 1. Lancet. 1994 Apr 2;343(8901):824-7. doi: 10.1016/s0140-6736(94)92026-5. PMID 7908078
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Background] Thiesmeier R, Orsini N. Rolling the DICE (Design, Interpret, Compute, Estimate): Interactive Learning of Biostatistics With Simulations. JMIR Med Educ. 2024 Apr 15;10:e52679. doi: 10.2196/52679. PMID 38619866
- [Background] Pezoulas VC, Zaridis DI, Mylona E, Androutsos C, Apostolidis K, Tachos NS, Fotiadis DI. Synthetic data generation methods in healthcare: A review on open-source tools and methods. Comput Struct Biotechnol J. 2024 Jul 9;23:2892-2910. doi: 10.1016/j.csbj.2024.07.005. eCollection 2024 Dec. PMID 39108677
- [Background] Zhang Z, Yan C, Mesa DA, Sun J, Malin BA. Ensuring electronic medical record simulation through better training, modeling, and evaluation. J Am Med Inform Assoc. 2020 Jan 1;27(1):99-108. doi: 10.1093/jamia/ocz161. PMID 31592533
- [Background] Sun C, Dumontier M. Generating unseen diseases patient data using ontology enhanced generative adversarial networks. NPJ Digit Med. 2025 Jan 3;8(1):4. doi: 10.1038/s41746-024-01421-0. PMID 39753917